CLINICAL TRIAL: NCT06215885
Title: Cancer Hospital Chinese Academy of Medical Sciences
Brief Title: Multi-omics Analysis to Characterize the Invasive Evolution of Pulmonary Subsolid Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC4258
Record Dates: First submitted 2024-01-01; First posted 2024-01-22 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of Lung
Keywords: Subsolid nodule; Invasive evolution
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subsolid nodules group: Patients with pulmonary subsolid nodules were identified by CT examination and intended for surgical treatment. All participants will undergo chest CT, genomic, and proteomic tests to identify related biomarkers and establish a clinical diagnostic model for the invasiveness of subsolid nodules.
  Interventions: Diagnostic Test: Mass spectrometry-based proteomics
- Volunteers group: Healthy volunteers.
  Interventions: Diagnostic Test: Mass spectrometry-based proteomics

INTERVENTIONS:
Diagnostic Test: Mass spectrometry-based proteomics — Detecting genomic and proteomic information
  Other Names: Phosphoproteomics; Deep-profiling tyrosine phosphorylation proteomics; Plasma proteomics; Plasma genomics; Whole-exome sequencing

SUMMARY:
Current clinical follow-up frequency and treatment timing for pulmonary subsolid nodules (SSNs) rely mostly on whether the nodules grow, which may not accurately reflect the pathological status, and may lead to unnecessary follow-ups. This study aims to use multi-omics techniques to dynamically observe the growth and invasiveness evolution process of SSNs and uncover its invasiveness mechanism. Radiological characteristics of SSNs in different invasiveness stages were also analyzed and summarized by analyzing preoperative CT. This can overcome the bottleneck of invasiveness assessment in the growth process of SSN and provide scientific evidence for the scientific management and clinical treatment timing choice of SSN patients, thus facilitating the rational allocation of medical resources and prolonging the expected survival of national health.

DETAILED DESCRIPTION:
This prospective observational cohort study aims to recruit 120 patients with subsolid nodules (SSNs) and 100 healthy volunteers. Enroll 120 patients with SSNs planned for surgery and 100 healthy volunteers. Sequence blood and tissue samples from patients and compare the relevance of biomarkers between the two. Use blood from healthy volunteers as blank controls. Additionally, analyzes radiological characteristics of SSNs at different invasive stages using preoperative CT.

ELIGIBILITY:
Inclusion Criteria:

Patients with SSNs

1. Newly diagnosed patients with persistent SSNs confirmed by thin-section chest CT examination
2. Patient areilling to undergo surgery
3. Voluntarily sign a written informed consent form

Healthy Volunteers

1. Healthy volunteers aged 18-50 years, regardless of gender.
2. No lung nodules detected on chest thin-section CT.
3. No history of cancer.
4. Voluntary sign a written informed consent form.

Exclusion Criteria:

Patients with SSNs

1. Surgical contraindications
2. Inability to cooperate with CT/MR examination to obtain high-quality images
3. History of malignant tumors
4. Previous targeted, immune, or ablation therapy
5. Postoperative pathology of non-lung adenocarcinoma disease spectrum
6. Other situations deemed unsuitable for participation in this study by the researchers

Healthy Volunteers

1. Drug abuse
2. HIV infection or AIDS
3. History of syphilis, gonorrhea, or other infectious diseases
4. Hepatitis B or C virus carrier

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent chest CT examination and found SSN and planned to undergo surgical treatment from November 2023 to September 2024 and Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of subsolid nodule invasive diagnosis | Through study completion, an average of 1 year.
  The efficacy of screening features for SSN invasiveness was compared to pathological diagnosis, using metrics such as sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No